CLINICAL TRIAL: NCT02669719
Title: A Randomized Phase II Study to Evaluate Efficacy and Safety of DCVAC/LuCa Added to Chemotherapy With Carboplatin and Pemetrexed vs Chemotherapy Alone in Patients With Stage IV Non-small Cell Lung Cancer
Brief Title: Cellular Immunotherapy Synergize Chemotherapy in Patients With Stage IV NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: SOTIO a.s. (Industry)
Responsible Party: Principal Investigator, Baohui Han, Vice-President, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILU02
Record Dates: First submitted 2016-01-11; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy followed dendritic cells (Experimental): pemetrexed and carboplatin chemotherapy followed dendritic cells infusion from Cycle 3
  Interventions: Biological: chemotherapy followed dendritic cells
- chemotherapy (Active Comparator): pemetrexed and carboplatin chemotherapy only
  Interventions: Drug: pemetrexed and carboplatin

INTERVENTIONS:
Biological: chemotherapy followed dendritic cells — Pemetrexed and carboplatin would be administered on day 1 of each 3-week cycle.Patients will start with dendritic cells treatment on Day 15 of pemetrexed and carboplatin chemotherapy from Cycle 3 provided that both leukapheresis and the production of dendritic cells are successful.
  Arms: chemotherapy followed dendritic cells
Drug: pemetrexed and carboplatin — Chemotherapy with 4-6 cycles of pemetrexed and carboplatin as first-line induction chemotherapy followed by pemetrexed as maintenance therapy.
  Arms: chemotherapy

SUMMARY:
This is a randomized, open-label, phaseⅡ study evaluating efficacy and safety of DC (dendritic cells) vaccine concurrent with chemotherapy compared to chemotherapy alone in patients with stage IV NSCLC (non small cell lung cancer) with wild-type EGFR (epidermal growth factor receptor).

DETAILED DESCRIPTION:
Screening period: Patients will be screened for eligibility for the clinical study within a 4-week period.

Randomization and leukapheresis periods: When the patients meet all entry criteria, they will be randomized in a ratio of 1:1 into one of the following two groups:

Group A (experimental group): Treatment with DC in addition to chemotherapy with 4-6 cycles of pemetrexed/carboplatin as first-line induction chemotherapy followed by pemetrexed as maintenance therapy. These patients will undergo leukapheresis within 1 week after randomization before start of treatment.

Group B (control group): Chemotherapy with 4-6 cycles of pemetrexed/carboplatin as first-line induction chemotherapy followed by pemetrexed as maintenance therapy.

Treatment periods:

Standard of care chemotherapy will be administered to patients in both treatment groups in cycles. Each chemotherapy cycle will be 3 weeks long. Patients in the group A will start with chemotherapy 2-5 days after leukapheresis, and patients in the group B will start with chemotherapy within 2 weeks after randomization.

Induction chemotherapy period

Pemetrexed in combination with carboplatin will be administered on Day 1 of each 3-week chemotherapy cycle. After 2 cycles of chemotherapy, tumor response will be evaluated according to RECIST v. 1.1. Patients with progressive disease or intolerance to chemotherapy will terminate study treatment but will be followed for survival. Patients with complete response, partial response, or stable disease will continue chemotherapy with carboplatin and pemetrexed for a total of 6 cycles . After at least a total of 4 cycles of chemotherapy, patients can be administered pemetrexed maintenance chemotherapy.

Maintenance chemotherapy period

During the Maintenance chemotherapy period, patients will receive pemetrexed of each 3-week chemotherapy cycle. Chemotherapy with pemetrexed will be administered in up to a total of 21 cycles or until disease progression or development of intolerance.

DCVAC

Patients in the group A will start with DC treatment on Day 15 of chemotherapy Cycle 3 provided.During the Induction chemotherapy period, DC will be administered on Day 15 of each subsequent 3-week chemotherapy cycle of chemotherapy. During the Maintenance chemotherapy period, DC will be administered on Day 15 of every other 3-week chemotherapy cycle.

Follow-up periods: Patients who complete or discontinue all study treatments after Cycle 3 before disease progression will undergo disease evaluation by CT scan every 3 months until progression of the disease.Patients who discontinue all study treatments before or at Cycle 2 for any reason or those who complete or discontinue all study treatments after Cycle 3 after disease progression will be followed up for survival. The survival data will be collected every 3 months by directly contacting the patient (or a relative/caretaker) by phone until death from any reason or termination of the study. The clinical study will be terminated when at least 45 PFS (progression-free survival) events have been reached, which is assumed to happen approximately 24 months after start of treatment of the first patient included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IV, non-squamous, wild-type EGFR,ALK-negative NSCLC
2. Signed ICF and ability to comply with this protocol
3. 18 years of age or older
4. ECOG performance status of 0-1
5. Patients must have measurable disease as defined by RECIST v. 1.1
6. Systematic treatment naive with respect to the currently diagnosed NSCLC
7. Patients must have recovered from toxicity of previous therapy. Recovery is defined as less than or equal to grade 2 toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (except alopecia).
8. Sufficient hematologic and organ function for leukapheresis and chemotherapy:

   * WBC equal to or higher than 4×10^9 /L
   * Neutrophil equal to or higher than 1.5×10^9 /L
   * PLT equal to or higher than 100×10^9 /L
   * Hemoglobin equal to or higher than9 g/dL (90 g/L)
   * Total bilirubin less than or equal to 1.5 times upper limit of normal (benign hereditary hyperbilirubinemias, eg, Gilbert's syndrome are permitted)
   * Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) should be less than or equal to 3 times upper limit of normal. ALP, AST, and ALT less than or equal to 5 times upper limit of normal is acceptable if liver has tumor involvement.
   * Creatinine clearance equal to or higher than 45 mL/min (calculated with the standard Cockcroft and Gault formula)
9. Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the treatment plus 3 months

Exclusion Criteria:

1. Known active/untreated CNS metastases
2. Any known primary immunodeficiency
3. Any preexisting medical condition requiring long term chronic steroid or immunosuppressive therapy
4. HIV positivity, hepatitis B and/or C infection, syphilis
5. Past or current history of malignant neoplasm other than lung carcinoma, except for adequately treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least five years
6. Patient's significant co-morbidities:

   * Cardiovascular diseases - unstable angina pectoris, uncontrolled hypertension, myocardial infarction or ventricular arrhythmia or stroke within a 6-month period before randomization, congestive heart failure or cardiac arrhythmia not controlled by treatment
   * Active severe infections or other severe medical condition
7. Participation in a clinical study using experimental therapy and immunotherapy,monoclonal antibodies within the last 4 weeks prior to study entry
8. Pregnant or breastfeeding woman
9. History of severe hypersensitivity to pemetrexed and carboplatin and their ingredients, and to DCVAC ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | the time from the date of randomization to the date of an event defined as the first progression or death due to any cause, whichever occurs first, up to 24 months
  randomization to the date of an event defined as the first progression or death due to any cause (institution of a new systemic anticancer treatment will also be considered as a progression event),whichever occurs first up to 24 months

SECONDARY OUTCOMES:
Safety parameters in terms of AE, laboratory abnormalities, and vital signs | through study completion, an average of 24 months
  adverse events [AEs], serious adverse events [SAEs], adverse events of special interest [AESIs], laboratory abnormalities, and vital signs
Overall Survival | From study treatment to death due to any cause, up to 24 months
Objective Response Rate | Objective Response Rate measured by RECIST criteria in ITT population, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided